CLINICAL TRIAL: NCT05593042
Title: Phase 2, Randomized, Double-blind Study to Evaluate Immunogenicity Superiority of a Booster Dose With an Omicron or a Trivalent Vaccine Compared to CoronaVac, in Adults Immunized With Different Vaccine Schedules Against SARS-CoV-2 in Chile
Brief Title: Immunogenicity Evaluation of Omicron Variant-based Vaccine and a Trivalent Vaccine in Adults Against COVID-19 in Chile
Acronym: CoronaVarCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-tonCOV-2001-CL
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Vaccines
Keywords: Clinical Trials; COVID-19; Inactivated Vaccine; Omicron Vaccine; Trivalent Vaccine
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine; SARS-CoV-2 inactivated vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A specialized company designed the randomization algorithm of vaccines (IRT algorithm). The algorithm was designed considering the vaccination schedule of the subjects and the number of subjects assigned to each center. Once randomized, each participant will be assigned to a treatment branch/group. Neither the personnel administering it nor the rest of the team nor the participant will know which product was administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Heterologous group receiving CoronaVac® (Active Comparator): General population that received two doses of CoronaVac® as a primary schedule of vaccination and two booster doses as part of the national vaccination schedule with mRNA or viral vector-based vaccines; and who receive a booster dose of CoronaVac®
  Interventions: Biological: CoronaVac®
- Heterologous group receiving Omicron vaccine (Experimental): General population that received two doses of CoronaVac® as a primary schedule of vaccination and two booster doses as part of the national vaccination schedule with mRNA or viral vector-based vaccines; and who receive a booster dose of Omicron vaccine
  Interventions: Biological: Omicron Vaccine
- Heterologous group receiving a trivalent vaccine (Experimental): General population that received two doses of CoronaVac® as a primary schedule of vaccination and two booster doses as part of the national vaccination schedule with mRNA or viral vector-based vaccines; and who receive a booster dose of trivalent vaccine
  Interventions: Biological: Trivalent Vaccine
- Homologous group receiving Omicron vaccine (Experimental): Participants of the CoronaVac03CL study who have received the primary regimen and two booster doses with CoronaVac® vaccine; and who receive a booster dose of Omicron vaccine
  Interventions: Biological: Omicron Vaccine
- Homologous group receiving a trivalent vaccine (Experimental): Participants of the CoronaVac03CL study who have received the primary regimen and two booster doses with CoronaVac® vaccine and who receive a booster dose of trivalent vaccine
  Interventions: Biological: Trivalent Vaccine

INTERVENTIONS:
Biological: CoronaVac® — The active ingredient is the SARS-CoV-2 virus (CZ02 strain, ancestral) grown in Vero cells and inactivated, in aluminum hydroxide. The vaccine is preservative-free, and it is packed in pre-load syringes (0.5 mL) with 600 SU/0.5mL of inactivated SARS-CoV-2.
  Other Names: Inactivated SARS-CoV-2 Vaccine (Vero Cells) - Sinovac
  Arms: Heterologous group receiving CoronaVac®
Biological: Omicron Vaccine — An experimental intervention consisting of a booster dose of an inactivated Omicron variant vaccine.
  The active ingredient is the SARS-CoV-2 virus (Omicron variant) grown in Vero cells and inactivated, in aluminum hydroxide. The vaccine is preservative-free, packed in a pre-load syringe, and contains one dose (0.5mL) of 1200 SU of inactivated SARS-CoV-2 Omicron variant.
  Arms: Heterologous group receiving Omicron vaccine; Homologous group receiving Omicron vaccine
Biological: Trivalent Vaccine — An experimental intervention consisting of a booster dose of an inactivated trivalent (CZ02 strain, ancestral, Delta, and Omicron variants) variant vaccine.
  The active ingredient is the SARS-CoV-2 virus (CZ02 strain, ancestral, Delta, and Omicron variants) grown in Vero cells and inactivated, in aluminum hydroxide. The vaccine is preservative-free, and it is packed in a pre-load syringe containing one dose (0.5mL) (1200 SU of inactivated SARS-CoV-2 WT, 1200 SU of inactivated SARS-CoV-2 Delta variant, and 1200 SU of inactivated SARS-CoV-2 Omicron variant).
  Arms: Heterologous group receiving a trivalent vaccine; Homologous group receiving a trivalent vaccine

SUMMARY:
Phase 2 clinical trial in adults previously vaccinated against SARS-CoV-2 in Chile with an initial schedule of two doses of CoronaVac® plus two booster doses with different vaccines. Subjects will randomly receive a third booster dose with Omicron, trivalent, or CoronaVac® vaccine. The humoral immunogenicity against COVID-19 will be compared in subjects that received the Omicron or the Trivalent vaccines with subjects that received CoronaVac® to determine the superiority of the two candidate vaccines versus CoronaVac®. Subjects will be followed for 6 months after the booster dose administration.

DETAILED DESCRIPTION:
This study will be a phase 2 randomized, double-blind, multicenter clinical trial in fully vaccinated adults, males, and females, who have previously received an initial schedule of two doses of CoronaVac® plus two booster doses with different vaccines against SARS-CoV-2 in Chile. Two groups of participants will be included: Heterologous group: subjects who had received two booster doses with mRNA or viral vector-based vaccine); and homologous group: subjects who have received two booster doses of CoronaVac® in a previous clinical trial (CoronaVac03CL).

Subjects of the heterologous group will randomly receive a booster dose with Omicron, trivalent, or CoronaVac® vaccine. On the other hand, subjects of the homologous group will randomly receive a booster dose of Omicron or trivalent vaccine.

The humoral immunogenicity against COVID-19 will be compared in subjects of the heterologous group that will receive Omicron or trivalent vaccine with subjects that will receive CoronaVac®, to determine the superiority of the two candidate vaccines versus CoronaVac®.

Subjects will be followed for 6 months after the booster dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Adults, male or female, over 18 years of age;
* Fully vaccinated against SARS-CoV-2 with two initial doses of CoronaVac® vaccine and that have received two booster doses of a different vaccine (heterologous group) or with CoronaVac® (homologous group) at least 5 months before enrollment;
* Capable of understanding and signing the informed consent form;
* Availability and commitment to comply with study procedures and in-person and remote appointments.

Exclusion Criteria:

* Symptomatic COVID-19 diagnosed 60 days before enrollment (confirmed COVID-19 by RT-PCR or antigen test, or by being in close contact with a confirmed case);
* Pregnant women (confirmed by urine pack test) or women who plan to get pregnant within the first 3 months of the study;
* Known allergies to the vaccine components;
* Evidence of uncontrolled metabolic, neurologic#, cardiac, pulmonary, hepatic, or renal disease. Significant changes in medical treatment or hospitalizations due to worsening conditions in the last three months are indicators of uncontrolled disease or unsuccessful adherence to the treatment;
* Alteration of the immune system (neoplasms, except basal cell cancer), congenital or acquired immunodeficiencies, and uncontrolled autoimmune diseases. Significant changes in medical treatment or hospitalizations due to worsening conditions in the last three months are indicators of uncontrolled disease;
* Behavioral, psychiatric, or cognitive conditions# that, according to the study physician, impair the ability to understand and cooperate with the requirements of this trial;
* Intake of immunosuppressants within 6 months before enrollment or prescribed to be taken within the next 2 years of the study. Antineoplastic therapy, radiation, and immunosuppressants that induce tolerance to transplants, among others, are included in this category;
* Intake of corticosteroids within 3 months before enrollment or prescribed to be taken within 3 months after enrollment. The equivalent of 20 mg/day of prednisone for more than one week will be considered an immunosuppressive dose. Topical or inhaled steroids are not considered immunosuppressive drugs;
* History of anatomic or functional asplenia;
* Coagulation disorders such as coagulation factor deficiency, coagulopathy or platelet disorders, or a history of significant bleeding or bruising from intramuscular injections or venipunctures;
* Alcohol or drug abuse reported 12 months before enrollment that caused medical, professional, or family consequences;
* Have been treated with blood or immunoglobulin transfusions within 3 months before enrollment;
* Have you received any live attenuated or inactivated vaccine within 28 and 14 days prior to the enrollment or planned to receive one within the first 28 days of the study;
* Participation in another clinical trial 6 months before the enrollment or plan to participate in one 6 months after the enrollment in this trial;
* Prior participation in a SARS-CoV-2 vaccine trial different than the CoronaVac03CL trial;
* Any fever episode (body temperature ≥37.8℃) within 3 days before enrollment;
* Any other condition that according to the primary care physician, could jeopardize the safety/rights of the subject or prevent him/her from completing the protocol

  * Alzheimer's and senile dementia are exclusion criteria.

Note: Obese and smoker participants are allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Superiority in humoral immunogenicity of the neutralizing antibodies against the Delta and Omicron variants in response to a booster dose of the trivalent vaccine compared to CoronaVac® in adults previously immunized against SARS-CoV-2. | Up until 6 months after intervention
  Differences in the humoral immunogenicity (GMT ratio >1) of the neutralizing antibodies against the Delta and Omicron variants in response to a booster dose of the trivalent vaccine compared to CoronaVac® in adults who have initially received two doses of CoronaVac® and two booster doses with vaccines against SARS-CoV-2 different from CoronaVac® (mRNA or viral vectors (heterologous group)) will be evaluated.
Superiority in humoral immunogenicity of neutralizing antibodies against the Omicron variant in response to a booster dose with the Omicron vaccine when compared with CoronaVac® in adults previously immunized against SARS-CoV-2. | Up until 6 months after intervention
  Differences in the humoral immunogenicity (GMT ratio >1) of the neutralizing antibodies against the Omicron variant generated in response to a booster dose with the Omicron vaccine when compared with CoronaVac® in adults who have initially received two doses of CoronaVac® and two booster doses with vaccines against SARS-CoV-2 different from CoronaVac® (mRNA or viral vectors (heterologous group)) will be evaluated.
Non-inferiority of neutralizing antibodies against the Omicron and Delta variants generated by a booster dose of trivalent vaccine when compared to CoronaVac® in adults previously immunized against SARS-CoV-2 in a heterologous schedule. | Up until 6 months after intervention
  Evaluation of the non-inferiority (seroconversion rate ≥5%) of neutralizing antibodies against the Omicron and Delta variants generated by a booster dose of trivalent vaccine when compared to CoronaVac® in adults who have initially received two doses of CoronaVac® and two booster doses with vaccines from other platforms (mRNA or viral vectors (heterologous group)).
Non-inferiority of neutralizing antibodies against the Omicron variant generated by a booster dose with Omicron vaccine when compared with CoronaVac® in adults previously immunized against SARS-CoV-2 in a heterologous schedule. | Up until 6 months after intervention
  Evaluation of the non-inferiority (seroconversion rate ≥5%) of neutralizing antibodies against the Omicron variant generated by a booster dose with Omicron vaccine when compared with CoronaVac® in adults who have two doses of CoronaVac® and two booster doses with vaccines from other platforms (mRNA or viral vectors (heterologous group)).

SECONDARY OUTCOMES:
Frequency of adverse events within the 7 and 28 days after the administration of a booster dose of Omicron, trivalent or CoronaVac® vaccines. | 28 days after intervention
  Evaluate whether there are differences in the frequency of adverse events within the 7 and 28 days after the administration of a booster dose of Omicron, trivalent or CoronaVac® vaccines.
Serious adverse events (SAE) and adverse events of special interest (AESI) in participants who received a booster dose of the Omicron, trivalent, or CoronaVac® vaccines. | Up until 6 months after intervention
  Follow up of serious adverse events (SAE) and adverse events of special interest (AESI) will be performed for participants who received a booster dose of the Omicron, trivalent, or CoronaVac® vaccines.
Humoral immunogenicity against the ancestral strain induced by a booster dose with Omicron vaccine or trivalent vaccine in adults previously immunized against SARS-CoV-2 in a heterologous schedule. | Up until 6 months after intervention
  Evaluation of the humoral immunogenicity (GMT and seroconversion rate of neutralizing antibodies) against the ancestral strain, induced by a booster dose with Omicron vaccine or trivalent vaccine in adults who have two doses of CoronaVac® and two booster doses with vaccines from other platforms (mRNA or viral vectors (heterologous group)).
Humoral immunogenicity induced by a booster dose with Omicron or trivalent vaccine in adults previously immunized against SARS-CoV-2 in a homologous schedule. | Up until 6 months after intervention
  To evaluate the humoral immunogenicity (GMT and seroconversion of neutralizing antibodies) induced by a booster dose with Omicron or trivalent vaccine in adults who have previously received four doses of CoronaVac® (homologous group) against the ancestral strain, the Omicron, and Delta variants.
Cellular immunogenicity generated, in a subgroup of participants, by the administration of a booster dose with Omicron, trivalent or CoronaVac® vaccines against the ancestral strain, the Omicron and Delta variants. | Up until 6 months after intervention
  To evaluate, in a subgroup of participants, the cellular immunogenicity (T cell activation and cytokines secretion) generated by the administration of a booster dose with Omicron, trivalent or CoronaVac® vaccines against the ancestral strain, the Omicron and Delta variants.
Levels of neutralizing antibodies -and in a subgroup of subjects, the cellular immunity- against the ancestral, Omicron and Delta strains at 6 months after the intervention. | 6 months after intervention
  Evaluation of the levels of neutralizing antibodies in every participant and the cellular immunity in a subgroup of subjects against the ancestral strain, the Omicron and Delta variants at 6 months after the administration of a booster dose of the Omicron, trivalent or CoronaVac® vaccines.

OTHER OUTCOMES:
The humoral and cellular immunogenicity, in a subgroup of participants (homologous and heterologous groups), against new variants of concerns identified during the development of this trial. | Up until 6 months after intervention
  The humoral and cellular immune response elicited against new variants of concerns identified during the development of this trial will be evaluated in a subgroup of participants (homologous and heterologous groups).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo A Gonzalez, PhD, Study Director — Pontificia Universidad Catolica de Chile; Alexis M Kalergis, PhD, Study Chair — Pontificia Universidad Catolica de Chile; Susan M Bueno, PhD, Study Chair — Pontificia Universidad Catolica de Chile; Katia Abarca, MD, Study Chair — Pontificia Universidad Catolica de Chile
Locations (3):
- Chile (3):
  - Universidad del Desarrollo - Clínica Alemana, Santiago, RM
  - Pontificia Universidad Católica - Marcoleta Center, Santiago, Santiago Metropolitan
  - Universidad San Sebastián, Santiago, Santiago Metropolitan

REFERENCES:
- [Derived] Mendez C, Rodriguez-Guilarte L, Palacios PA, Gutierrez-Vera C, Roman F, Moreno-Tapia D, Rios M, Reyes A, Cancino FA, Otero FF, Zurita C, Rivera D, Cabrera A, Duarte LF, Urzua M, Iturriaga C, Rojas A, Perez CM, Redlich AS, Fasce RA, Fernandez J, Mora J, Ramirez E, Dominguez A, Weiskopf D, Grifoni A, Sette A, Zeng G, Meng W, Goldbatt D, Johnson M; CoronaVarCL study group; Gonzalez-Aramundiz JV, Alvarez-Figueroa MJ, Abarca K, Carreno LJ, Gonzalez PA, Kalergis AM, Penaloza HF, Bueno SM. A booster dose of an inactivated SARS-CoV-2 vaccine targeting virus variants sustains protective humoral and cellular immunity. BMC Med. 2025 Dec 15. doi: 10.1186/s12916-025-04535-8. Online ahead of print. PMID 41398275